CLINICAL TRIAL: NCT06496113
Title: Recurrence ad Survival After Robotic Versus Laparoscopic Liver Resection in Very-early to Early (BCLC 0-A) Hepatocellular Carcinoma
Brief Title: Robotic Versus Laparoscopic Liver Resection for Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-01022 CE 4377
Record Dates: First submitted 2024-07-01; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robotic liver resections
  Interventions: Procedure: Minimally invasive liver resection
- Laparoscopic liver resection
  Interventions: Procedure: Minimally invasive liver resection

INTERVENTIONS:
Procedure: Minimally invasive liver resection — Patients underwent liver resection either by robotic or laparoscopic approach

SUMMARY:
The objective of the study is to investigate the long-term outcomes of minimally invasive liver surgery (robotic vs laparoscopic) for hepatocellular carcinoma patients of stage BCLC 0-A. Data from two tertiary centers for liver surgery will be retrospectively reviewed. Patients will be divided in two cohorts (robot; laparoscopy). The primary endpoint will be recurrence-free and overall survival; secondary endpoints were incidence, pattern, and treatment of recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing robotic and laparoscopic resections
* Histology-confirmed HCC of stage BCLC 0-A
* Preserved liver function (Child score A-B)
* Patients >18 years old

Exclusion Criteria:

* Hand-assisted procedures
* Non-elective surgery
* Intraoperative switch to locoregional therapies (like radiofrequency or microwave ablation)
* Non-histologically confirmed HCC
* Mixed hepato-cholangiocarcinoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients underwent minimally invasive liver resection in centers participating in the study
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2024-04 (Actual); Study Completion 2024-06 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival | From the date of liver resection until the first documented HCC progression on follow-up imaging, assessed up to 116 months. The Minimum follow-up accepted was of 3 months postoperatively.
  Recurrence was dated at the first HCC detection on follow-up imaging.
Overall survival | From the date of liver resection until the date of death for any cause or the last follow-up available whichever came first, assessed up to 116 months. The Minimum follow-up accepted was of 3 months postoperatively.